CLINICAL TRIAL: NCT03024957
Title: Effect of Intrathecal Morphine, Dexmedetomidine or Both in Combination to Bupivacaine on Immunity in Patients Undergoing Major Abdominal Cancer Surgeries
Brief Title: Effect of Intrathecal Morphine, Dexmedetomidine or Both in Combination to Bupivacaine on Immunity
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Shereen Mamdouh, Lecturer of anesthesia, ICU and pain managment, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 123
Record Dates: First submitted 2017-01-11; First posted 2017-01-19 (Estimated); Last update posted 2021-01-14 (Actual); Status verified 2021-01

CONDITIONS: Immune System Suppression
Keywords: morphine; dexmedetomidine; immune system
MeSH Terms: interventions — Morphine; Dexmedetomidine; Bupivacaine

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Dexmedetomidine group (Active Comparator): patients received 10 mg of hyperbaric bupivacaine 0.5% in 2 mL volume and 5 μg of dexmedetomidine in 1 mL volume intrathecally.
  Interventions: Drug: Dexmedetomidine; Drug: Bupivacaine
- Morphine group (Active Comparator): patients received 10 mg of hyperbaric bupivacaine 0.5% in 2 mL volume and 0.5 mg morphine sulphate in 1 mL volume intrathecally.
  Interventions: Drug: Morphine Sulfate; Drug: Bupivacaine
- Dexmedetomidine + morphine group (Active Comparator): patients received 10 mg of hyperbaric bupivacaine 0.5% in 2 mL volume and 5 μg of dexmedetomidine plus 0.5 mg of morphine sulphate in 1 mL volume intrathecally.
  Interventions: Drug: Morphine Sulfate; Drug: Dexmedetomidine; Drug: Bupivacaine

INTERVENTIONS:
Drug: Morphine Sulfate — Intrathecal injection as the patients will be placed in the sitting position and a 25-gauge Quincke needle will be placed in the L2-3 or L3-4 interspaces with injection of morphine sulphate .
  Arms: Dexmedetomidine + morphine group; Morphine group
Drug: Dexmedetomidine — Intrathecal injection as the patients will be placed in the sitting position and a 25-gauge Quincke needle will be placed in the L2-3 or L3-4 interspaces.
  Arms: Dexmedetomidine + morphine group; Dexmedetomidine group
Drug: Bupivacaine — Intrathecal injection as the patients will be placed in the sitting position and a 25-gauge Quincke needle will be placed in the L2-3 or L3-4 interspaces.

SUMMARY:
this work aims to investigate the effect of intrathecal administration of Morphine, Dexmedetomidine or both in combination on cellular immunity and cytokine production in patients undergoing major abdominal cancer surgeries.

DETAILED DESCRIPTION:
Intrathecal (IT) adjuvants prolong the duration of spinal anesthesia and postoperative analgesia thereby reducing the requirement of postoperative supplemental analgesics. The incorporation of adjuvants also lowers the overall dose of local anesthetic and hence associated side effects. Morphine has been used widely to alleviate various types of pain and to supplement general anesthesia. On the other hand, morphine has been reported to possess some immunosuppressive effects. Postoperative immunity is also important in conjunction with defence against malignant tumour. Dexmedetomidine is a highly selective α2 agonist with analgesia, sedation, anxiolysis, and sympatholysis as its useful pharmacological actions. The extended analgesic efficacy of IT dexmedetomidine (ITD) in the postoperative period has been shown in a few clinical studies. In addition, current insights have identified that dexmedetomidine has a capacity in inhibiting the overproduction of a variety of inflammatory molecules including TNF-α, IL-1β, and IL-6 in several acute inflammatory animal models.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II patients scheduled for major abdominal cancer surgeries

Exclusion Criteria:

* patients with known allergy to the study drugs,
* significant cardiac, respiratory, renal or hepatic disease,
* drug or alcohol abuse,
* psychiatric illness that would interfere with perception and assessment of pain.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-01; Primary Completion 2018-09 (Actual); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
Change from the base line in cellular immunity | Baseline , immediate postoperative, 4 hours postoperative and 24 hours postoperative
  CD3, CD4, CD4/CD8, CD16, CD56

SECONDARY OUTCOMES:
Change from baseline in Cytokines | Baseline, immediate postoperative, 4 hours postoperative and 24 hours postoperative
  interleukin-1B, interleukin-6, interleukin-10 and tumor necrosis factor

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No